CLINICAL TRIAL: NCT04791098
Title: Impact of Infectious Diseases Consultation on Vaccination Coverage Among People Waiting for a Kidney Transplant at the Clermont-Ferrand Hospital
Acronym: PREVAGREF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2019 LESENS; 2019-A02304-53 (Other: ANSM)
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Kidney Transplantation
Keywords: Immunization Coverage; Transplant Recipient; Transplantation, Kidney; Infectious Disease Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stronger pre-transplant check-up (Experimental): routine patient management + specific infectious diseases consultation
  Interventions: Other: Specific infectious diseases consultation
- Standard pre-transplant check-up (No Intervention): routine patient management + letter sent to nephrologist

INTERVENTIONS:
Other: Specific infectious diseases consultation — Specific infectious diseases consultation at Clermont Ferrand Hospital with a specialist doctor :
  * Update vaccinations
  * Advice to travelers
  * Diagnostic and treatment of latent tuberculosis infection
  Arms: Stronger pre-transplant check-up

SUMMARY:
Solid-organ transplant patients are at increased risk of infectious diseases. Among this population, infectious diseases may be life-threatening or lead to graft rejection. Their prevention is an important challenge. Despite specific national recommendations, vaccination is underutilized. That is why we propose a dedicated infectious diseases consultation during pre-kidney transplantation assessment.

DETAILED DESCRIPTION:
The main objective of this study is to impove vaccine coverage before kidney transplantation.

Enrollment was based on the waiting list for a kidney transplant. Patients newly listed are invited to participate by the transplant team (nephrology department) ; for those that are already registered, a notification letter is sent to their home.

All patients included must :

* complete a health questionnaire
* take a blood test at day 0 : viral, bacterial and parasitic serologies, QuantiFERON-TB
* take a chest X-ray and dental panoramic Patients randomized in interventional group will be seen in specific infectious diseases consultation at Clermont Ferrand Hospital. A letter of recommendations is sent to nephrologist for patients randomized in group control.

The primary study endpoint (immunization coverage) is evaluated at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* On the waiting list for kidney transplantation at Clermont-Ferrand
* Free and informed consent
* Affiliation to a social security system

Exclusion Criteria:

* Patient under 18
* Protected adults (individuals under guardianship by court order
* Pregnant and nursing women
* Prior graft (solid organs or hematopoietic stem cells)
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Vaccination coverage | Month 6
  The percentage of fully immunized patients according to the Recommendations of High Council for public Health

SECONDARY OUTCOMES:
Infectious complications | within the 6 months of the transplantation
  Infectious diseases which require special management (hospitalization, anti-infective treatments)
Mortality | Month 6
  Mortality after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lesens, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France